CLINICAL TRIAL: NCT06574425
Title: A Multicenter, Prospective, Cohort Study on the Safety and Efficacy of Long-term, High Blood Flow Hemoadsorption Therapy in Patients Undergoing Maintenance Hemodialysis
Brief Title: Long-term, High Blood Flow Hemoadsorption Therapy in Patients Undergoing Maintenance Hemodialysis
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Dongliang Zhang, MD (Other)
Responsible Party: Sponsor-Investigator, Dongliang Zhang, MD, Director of Nephrology Department of Beijing Jishuitan Hospital, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2024081208
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Chronic Kidney Diseases; Hemodialysis
Keywords: protein-bound uremic toxins; hemoadsorption
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing maintenance hemodialysis with once-weekly hemoadsorption (Experimental): The blood flow rate is based on the actual blood flow speed displayed by the dialysis machine; the dialysis fluid flow rate is 500 ml/min; the total ultrafiltration volume in 4 hours does not exceed 4500 ml.All subjects undergo a self-controlled before-and-after comparison, with continuous 3 weeks of HA+HD treatment, once a week. The HA+HD treatment is implemented at a short interval of 1 day after the previous dialysis treatment. Group 1 is the routine treatment group, Group 2 is the extended time group, and Group 3 is the extended time and increased blood flow group, also known as the modified HA+HD group. The treatment modes of the three groups are implemented sequentially in order.
  Interventions: Other: long-term, high blood flow hemoadsorption therapy

INTERVENTIONS:
Other: long-term, high blood flow hemoadsorption therapy — Group 1 is the routine treatment group, Group 2 is the extended time group, and Group 3 is the extended time and increased blood flow group

SUMMARY:
Objective：The purpose of the study is to confirm that extending the duration of hemoadsorption (HA) and increasing blood flow during the HA+hemodialysis (HD) treatment process is safe and feasible, and to verify that extending the HP treatment duration can further increase the clearance of protein-bound uremic toxins.

Methods: The study employs a multicenter, prospective, cohort design with a self-controlled before-and-after comparison. The duration of HA+HD treatment for maintenance hemodialysis (MHD) patients is extended to 4 hours, and the extracorporeal blood flow rate is increased to over 250-350 ml/min. The safety of the treatment is assessed by evaluating the safety of the procedure; the levels of relevant toxins in the patients' blood are measured before and after treatment, and the clearance rate of uremic toxins after a single treatment is calculated and compared with the self-controlled before-and-after data to determine whether the modified protocol can remove more uremic toxins.

ELIGIBILITY:
Inclusion Criteria:

Maintenance Hemodialysis Patients with Uremia receive regular HA+HD treatment

Exclusion Criteria:

Plasma albumin <30g/L, severe malnutrition or cachectic state; platelet count <40×10^9/L or >300×10^9/L; hypercoagulable state allergy to the hemoperfusion device; new cardiovascular or cerebrovascular diseases; poor vascular access function, extracorporeal circulation blood flow unable to reach 250ml/min ultrafiltration volume >4500ml in a single dialysis session use of non-heparin anticoagulants inability to comply with the procedures of this study other conditions deemed unsuitable for participation in this study by the investigator

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
protein-bound toxins | 1month
  the clearance of protein-bound toxins will change

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Department of Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China